CLINICAL TRIAL: NCT03301545
Title: The Metabolic Impact of Bariatric Surgery Compared to Best Diabetic Care on Manitoba's Urban Indigenous Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS20519 (B2017:023)
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Type2 Diabetes Mellitus; Obesity; Bariatric Surgery Candidate
Keywords: Bariatric surgery; Obesity; Type 2 Diabetes Mellitus; Indigenous Population; Randomized Control Trial; Glycoslyated Hemoglobin A1C; Anthropometric measurements; Medication Use
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Patients consenting to participate will be randomized to one of two groups: (1) fast-track to bariatric surgery, or (2) Best diabetic care under the guidance of an endocrinologist for one year. Note: participants in the best diabetic care group will have the option to undergo bariatric surgery after one year if desired.
Who Masked: Outcomes Assessor
Masking Description: Each study participant will be assigned a unique study identification number (study ID). All information/data regarding the participant will be collected using the Study ID. In this way, data analyses by the outcomes assessor will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fast-Track to Bariatric Surgery (Active Comparator): Patients will undergo standard of care for bariatric surgery patients in Manitoba and receive preoperative evaluation by the Centre for Metabolic and Bariatric Surgery (CMBS) team of nurses, dietitians, psychologist, and kinesiologist. Patients must attend the standard appointments and achieve the personalized program goals to be approved for laparoscopic Roux-En-Y gastric bypass surgery. Once approved, one of four surgeons performs surgery (within 12 months of randomization). Patients are followed post-operatively (by surgeon) at 6 weeks, and at 6 and 12 months. Pharmacologic glycemic control will be determined by an endocrinologist as per a standardized post-operative protocol. Post-procedural multidisciplinary follow-up occurs based on established CMBS guidelines (phone call 1 week post-operatively and an appointment at 3 and 12 months). Patients receive surgery within the current publically funded bariatric surgery program; no additional direct costs incurred by the patients.
  Interventions: Procedure: Fast-Track to Bariatric Surgery
- Best Diabetic Care Group (No Intervention): Patients will receive the best available medical practice for the treatment, education, and follow-up T2DM based on Manitoba Diabetes Care Recommendations and Diabetes Canada's clinical practice guidelines. Patients will have access to a general physician, endocrinologist, and a diabetes education nurse. An Endocrinologist will deliver the program to patients. Diabetes care, education and self-management support services will be provided by the Victoria General Hospital (VGH) Diabetes Education Centre; led by a registered nurse and dietitian. Patients will undergo individual diabetes management instruction which may include counseling on topics such as diet, exercise, smoking cessation, medications, diabetic complications, and blood sugar testing. Medical therapies, including pharmaceutical agents, will be determined on an individual basis as per standard protocol. There will be no direct patient-related medication costs (publicly funded).
- Retrospective Cohort (No Intervention): A retrospective cohort of non-Indigenous bariatric surgery patients from the Centre for Metabolic and Bariatric Surgery Program will allow comparison with the intervention group. The cohort will be age and gender matched.

INTERVENTIONS:
Procedure: Fast-Track to Bariatric Surgery — 30 participants from the urban Indigenous community who have Type 2 diabetes and are candidates for bariatric surgery at the Centre for Metabolic and Bariatric Surgery will be randomized to the fast-track to bariatric surgery group.
  Arms: Fast-Track to Bariatric Surgery

SUMMARY:
Obesity and type 2 diabetes mellitus (T2DM) are major global health concerns as they commonly co-occur and are associated with significant morbidity, mortality, and health care expenditures. The Indigenous (First Nations, Metis and Inuit) population bears a disproportionate burden of T2DM in Canada. The prevalence of obesity among Indigenous individuals is approximately 31.2% compared to 18.6% for the non-Indigenous population. In 2011, 16.7% of Manitoba's population, or four times the Canadian average, identified as Indigenous. At the same time, prevalence of T2DM in Manitoba is on the rise. Bariatric surgery is an effective treatment modality for the improvement and resolution of T2DM in patients who are obese. We aim to compare the effectiveness of bariatric surgery with conventional medical treatment in treating metabolic diseases in Indigenous people; the findings of which will assist in future treatment and program planning. Our objective is to determine whether Manitoba's urban Indigenous population will achieve better diabetic control and improved rates of remission of T2DM with bariatric surgery compared to best diabetic medical care.

DETAILED DESCRIPTION:
Obesity and type 2 diabetes mellitus (T2DM) are major global health concerns as they commonly co-occur and are associated with significant morbidity, mortality, and health care expenditures. The Indigenous population bears a disproportionate burden of T2DM in Canada. The 2007/2008 Canadian Community Health Survey (Statistics Canada) reported the prevalence of obesity among Indigenous individuals is approximately 31.2% compared to 18.6% for the non-Indigenous population. In 2011, 16.7% of Manitoba's population, or four times the Canadian average, identified as Indigenous (Statistics Canada). At the same time, prevalence of T2DM in Manitoba is on the rise. Bariatric surgery is an effective treatment modality for the improvement and resolution of T2DM in patients who are obese. To date, there are no published studies comparing the effectiveness of bariatric surgery with conventional medical treatment in treating metabolic diseases in Indigenous people.

Our objective is to determine whether Manitoba's urban Indigenous population will achieve better diabetic control and improved rates of remission of T2DM with bariatric surgery compared to best diabetic medical care (Manitoba Diabetes Care Recommendations, 2010; consistent with the Diabetes Canada and Clinical Practice Guidelines). Our primary outcome is best diabetic control at one-year post-intervention, as measured by fasting plasma glucose and hemaglobin A1c (HbA1c). Secondary outcomes will include changes in diabetic medication use, mean weight loss, and percentage changes in blood pressure, waist circumference measurement changes, and levels of fasting blood lipids (total cholesterol, HDL, LDL, and triglycerides). Additional funding to extend the study to include follow-up of study participants at five years post-treatment through accessing their medical charts and anonymized administrative data will be sought.

ELIGIBILITY:
Inclusion Criteria:

* Urban Indigenous patient
* 18 to 55 years of age
* male of female
* Body Mass Index = or > 35 to 55 Kg/m2
* Confirmed diagnosis of Type II diabetes mellitus (HbA1c of 7.0% for at least one year)
* Referred and accepted as into the Centre for Metabolic and Bariatric Surgery Program

Exclusion Criteria:

* Currently a smoker
* Body Mass Index above 55 Kg/m2
* Diagnosed with Type I diabetes mellitus
* Have had previous bariatric surgery
* Have contraindications to laparoscopic and/or bariatric surgery
* Rural patients; due to lack of rural Indigenous community-based support necessary for bariatric surgery

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Fasting Blood Glucose | Baseline,3, 6, 9, and 12 months for all patients
  Change from baseline fasting blood glucose level at 3, 6, 9, and 12 months
Change in Glycosylated Hemoglobin (HbA1c) | Baseline,3, 6, 9, and 12 months for all patients
  Change from baseline Glycosylated Hemoglobin (HbA1c) at 3, 6, 9, and 12 months

SECONDARY OUTCOMES:
Change in Diabetic Medication | Baseline,3, 6, 9, and 12 months for all patients
  Change from baseline in the number and dose of diabetic medication at 3, 6, 9, and 12 months
Change in Mean Weight Loss | Baseline, at 3, 6, 9, and 12 months for all patients
  Change from baseline in total amount of weight lost at 3, 6, 9, and 12 months
Change in the Percentage Change in Blood Pressure | Baseline, at 3, 6, 9, and 12 months for all patients
  Change in Blood Pressure (percentage of initial pre-surgery blood pressure) at 3, 6, 9, and 12 months
Change in Waist Circumference | Baseline, at 3, 6, 9, and 12 months for all patients
  Change in waist circumference (cm) from baseline at 3, 6, 9, and 12 months
Change in Fasting Blood Lipids | Baseline, at 3, 6, 9, and 12 months for all patients
  Change in total, LDL, HDL, and triacylglycerides from baseline at 3, 6, 9, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Krista M Hardy, MD, Principal Investigator — University of Manitoba; Dept of Surgery

IPD SHARING:
Plan to Share IPD: Undecided
Will be carried out according to University of Manitoba and Winnipeg Regional Health Authority applicable policies.